CLINICAL TRIAL: NCT05889975
Title: The Efficacy of Different Adjunctive Plaque Control Modalities in Orthodontic Patients: a 30 Days Randomized Clinical Trial
Brief Title: The Efficacy of Different Adjunctive Plaque Control Modalities in Orthodontic Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Baghdad (Other)
Responsible Party: Principal Investigator, Ola Issam Majeed Aljanabi, Principal Investigator, University of Baghdad
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 738622
Record Dates: First submitted 2023-05-11; First posted 2023-06-05 (Actual); Last update posted 2024-07-08 (Actual); Status verified 2024-07

CONDITIONS: Gingivitis
Keywords: Dental plaque; Interdental brush; Single tufted brush; Water irrigator
MeSH Terms: conditions — Gingivitis; Dental Plaque

STUDY DESIGN:
Who Masked: Investigator
Masking Description: the examiner will be blinded to type of intervention given to the participants. Each intervention will be given a code which will be concealed by a third-party who have no role in the study. The codes will be declared at the end of the study during data analysis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- interdental tooth brush (Active Comparator): the patients will be instructed to brush their teeth for 2 minutes with a pea- size amount of dentifrice twice daily,then the brush will be used after completion of manual tooth brushing it will be gently inserted between the teeth and orthodontic appliance, the patient will be instructed to use appropriate size brush and a smaller brush size if it feels too tight.
  Interventions: Device: interdental brush
- single tufted brush (Active Comparator): the patients will be instructed to brush their teeth for 2 minutes with a pea- size amount of dentifrice twice daily,then the brush will be used after completion of manual tooth brushing it will be gently inserted between the teeth and orthodontic appliance.
  Interventions: Device: single tufted brush
- water irrigator (Active Comparator): the patients will be instructed to brush their teeth for 2 minutes with a pea- size amount of dentifrice twice daily,thenThe patients will be instructed to use water irrigator after manual tooth brushing with 300ml distal water placed in its container. The patients instructed to use the entire 300ml during each irrigation.
  Interventions: Device: water irrigator

INTERVENTIONS:
Device: interdental brush — cleaning the inter dental areas after manual tooth brush twice daily by the patient for 30 days
  Arms: interdental tooth brush
Device: single tufted brush — cleaning the inter dental areas after manual tooth brush twice daily by the patient for 30 days
  Arms: single tufted brush
Device: water irrigator — using water irrigator after manual tooth brushing twice daily with 300ml distal water placed in its container. The patients instructed to use the entire 300ml during each irrigation for 30 days
  Arms: water irrigator

SUMMARY:
Bacterial plaque is the primary etiological factor for periodontal disease ranging from mild gingival inflammation to severe periodontitis.The fixed appliance can alter the microbial composition of the oral environment.Patients who wear fixed braces must perform optimum oral hygiene techniques .using a regular toothbrush alone for plaque removal is important but it is not adequate;therefore,an Adjunctive Plaque Control such as inter dental brush ,single tufted brush and water irrigator are helpful.the objective of this study To compare the efficacy of water irrigator ,single tufted and interdental brush in reducing gingival inflammation and plaque accumulation and To determine the profile of the salivary (MIF) at base line visit and after 4 weeks of the study .

DETAILED DESCRIPTION:
Bacterial plaque has been widely demonstrated to be the primary etiological factor for periodontal disease ranging from mild gingival inflammation to severe periodontitis .

The fixed appliance can alter the microbial composition of the oral environment, promoting bacterial plaque retention, decreasing self-cleaning skills, and causing gingival infection or enamel decalcification, as well as white spot lesions with soft-tissue recession and tooth abrasion.Patients who wear fixed braces must perform optimum oral hygiene techniques to avoid a variety of problems, including as caries, enamel demineralization, gingivitis, gingival hyperplasia, and periodontitis .

Plaque removal using a toothbrush is an efficient way to prevent decalcification. However, it is unclear whether using a regular toothbrush alone is adequate for plaque removal. Some authorities have suggested for the use of interdental/interspace brushes to eliminate plaque from 'hard to reach' places .There is some evidence show that interdental brushes decrease plaque in interdental regions in patients with pocketing, interdental spaces, and bridges. However; interspace and interdental brushes are small-headed toothbrushes with bristles that can clean small regions that standard toothbrushes cannot reach.

The removal of plaque has been proven to be safe and efficient with water flossers, as reported by the American Dental Association (ADA). A water flosser can also minimize gingivitis.Single-tufted toothbrushes are suggested for cleaning free surfaces and parts of the teeth that are difficult to reach with other oral hygiene tools.

ELIGIBILITY:
Inclusion Criteria:

* patients wearing fixed stainless steel orthodontic appliances in upper and lower jaw aving minimum of 20 teeth
* non-smoker with no history of any systemic disease and patients
* did not receive medical treatment in the last three months prior to the examination and sampling.

Exclusion Criteria:

* Patients with other type of orthodontic appliance rather than fixed appliance or patients having dental crowns or bridges
* handicapped patient or patients with limited manual dexterities
* pregnant or lactating women
* periodontitis patient
* patients unwilling to participate in study

Ages: 14 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 60 (Actual)
Dates: Start 2023-01-09 (Actual); Primary Completion 2023-04-08 (Actual); Study Completion 2023-06-05 (Actual)

PRIMARY OUTCOMES:
Change in BOP score | 0-30 Days
  For recording BOP score, the periodontal probe was inserted with gentle force into the sulcus/pocket until minimal resistance was felt. The probing force presumably was ranging between 20 to 25g. The examination started from the distal surface of the right upper 7 moving mesially to measure all the existing teeth. For each tooth, 6 surfaces were examined; the surface that displayed bleeding on probing was scored 1 and the surface with no bleeding was scored 0
change in Gingival index | 0 -30 Days
  Subjects will undergo the measurement of gingival index according to Loe & Silness, designed to assess the severity and quality of gingival inflammation in an individual or population. The gingival inflammation is assessed on the basis of color, consistency and bleeding on probing. The gingiva surrounding the tooth is assessed at four sites: mesio-facial papilla, facial marginal gingiva, disto-facial papilla and lingual marginal gingiva. Data will be collected based on four possible clinical conditions: 0=Normal gingiva1=Mild Inflammation-Slight change in color, Slight odema. No bleeding on probing2=Moderate inflammation-redness,odema and glazing. Bleeding on probing 3=Sever inflammation-marked redness and edema.Ulceration.Tendency to spontaneous bleeding.
change in plaque index | 0-30 days
  Mean amount plaque between different comparators. Mean amount plaque between different comparators as anti-plaque agent after rinsing with different comparators using means of modified quigely hein plaque index[ Turesky ,1970

SECONDARY OUTCOMES:
Mean relative change in macrophage migration inhibition level in salivary Fluid | 0-30 days
  Mean relative change in macrophage migration inhibition level in salivary Fluid after brashing with different comparators from baseline at 30 days

CONTACTS AND LOCATIONS:
Locations (1):
- Ola, Baghdad, Iraq

IPD SHARING:
Plan to Share IPD: Undecided